CLINICAL TRIAL: NCT02125591
Title: Cranial-nerve Non-invasive Neuromodulation (CN-NINM) for Balance Deficits After Mild Traumatic Brain Injury: A Randomized, Double-Blinded, Sham-Controlled, Prospective Trial
Brief Title: Cranial-nerve Non-invasive Neuromodulation (CN-NINM) for Balance Deficits After Mild Traumatic Brain Injury (Full Trial)
Acronym: CN-NINM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); US Department of Veterans Affairs (U.S. Federal Agency); The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN-NINM full
Record Dates: First submitted 2014-04-07; First posted 2014-04-29 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2014-10

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active PoNS CN-NINM (Experimental): Active CN-NINM PoNS - Active cranial-nerve non-invasive neuromodulation (CN-NINM) using the Portable Neuromodulation Stimulator (PoNS) and balance/gait rehabilitation with physical therapy
  Interventions: Device: Active CN-NINM PoNS
- Sham PoNS CN-NINM (Sham Comparator): Sham CN-NINM PoNS - Sham cranial-nerve non-invasive neuromodulation (CN-NINM) using the Portable Neuromodulation Stimulator (PoNS) and balance/gait rehabilitation with physical therapy
  Interventions: Device: Sham CN-NINM PoNS

INTERVENTIONS:
Device: Active CN-NINM PoNS — Delivery of active stimulation of the tongue during in-person therapy sessions (1 hour) and during two home sessions (40 minutes) daily on 6 of 7 days per week (120 total sessions). Stimulation sessions will be separated by at least 4 hours.
  Other Names: Active cranial-nerve non-invasive neuromodulation (CN-NINM); Portable Neuromodulation Stimulator (PoNS)
  Arms: Active PoNS CN-NINM
Device: Sham CN-NINM PoNS — Delivery of sham stimulation of the tongue during in-person therapy sessions (1 hour) and during two home sessions (40 minutes) daily on 6 of 7 days per week (120 total sessions). Stimulation sessions will be separated by at least 4 hours.
  Arms: Sham PoNS CN-NINM

SUMMARY:
The purpose of this study is to evaluate improvement in balance after receiving physical therapy when augmented by CN-NINM than when augmented by a placebo (sham CN-NINM).

ELIGIBILITY:
Inclusion Criteria:

1. Veteran or Servicemember
2. 18 to 50 years old
3. Sustained one or more mild traumatic brain injury (mTBI)s
4. Demonstration of balance deficits on the Sensory Organization Test (a composite score of 75 or less (1/3 sample) and 72 or less (2/3 sample))
5. Available for the duration of the study

Exclusion Criteria:

1. History of traumatic brain injury (TBI) of any severity other than mild TBI
2. Presence of active substance abuse condition
3. Any condition for which posturography is contraindicated (e.g. leg amputation or fracture)
4. Diagnosed neurological disorder with balance sequelae, other than TBI (e.g. Parkinson's disease, incomplete spinal cord injury, or Multiple Sclerosis)
5. Orthostatic hypotension as defined by:

   1. A systolic blood pressure decrease (from supine to sitting) of at least 20 mmHg
   2. A diastolic blood pressure decrease of at least 10 mmHg, or
   3. A pulse increase of 30 beats or more per minute with associated signs or symptoms of cerebral hypoperfusion
6. An implanted medical device
7. Pregnancy
8. Oral infection
9. Known transmissible disease (HIV, hepatitis, influenza, TB)
10. Exam signs of serious disorder other than mTBI as defined by facial asymmetry, hoarseness and dysarthria (e.g. tumor, stroke).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Sensory Organization Test (SOT) | 12 weeks
  Comparison of the SOT score between the treatment group and sham group at the intermediate follow-up.

SECONDARY OUTCOMES:
Change in post-concussive symptoms using Neurobehavioral Symptom Inventory (NSI) | 12 weeks
Change in dizziness and unsteadiness measured by Dizziness Handicap Inventory (DHI) | 12 weeks
Change in space and motion discomfort measured by Situational Characteristics Questionnaire (SitQ) | 12 weeks
Change in quality of life measured using Short Form 36 (SF-36) | 12 weeks
Change in symptoms of post-traumatic stress disorder (PTSD) measured using the unspecified PTSD checklist (PCL-C) | 12 weeks
Change on neural organization in tracts controlling balance using diffusion tensor imaging (DTI) | 12 weeks
  DTI will be acquired using 3.0T field strength Siemens Trio MRI scanner.
Change in neuroimaging using functional magnetic resonance imaging (fMRI) | 12 weeks
  For fMRI, a repeated single-shot echo-planar imaging will be acquired

CONTACTS AND LOCATIONS:
Overall Officials: David X Cifu, MD, Principal Investigator — VA Department of Physical Medicine and Rehabilitation; William C Walker, MD, Principal Investigator — Virginia Commonwealth University (VCU)
Locations (2):
- United States (2):
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia